CLINICAL TRIAL: NCT07289399
Title: Is There a Benefit From Addition of Treadmill Walking to Diet Restriction in Psoriasis Women With PCOS?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Cardiovascular, Respiratory disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00014233-58
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Psoriasis; Polycystic Ovary Syndrome
MeSH Terms: conditions — Psoriasis; Polycystic Ovary Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): Group I will enroll twenty females with PCOS and Psoriasis who will apply forty minutes walking on treadmill three times per week. Also Group I will follow low calorie diet and daily metformin for 12 weeks.
  Interventions: Behavioral: exercise and diet restriction
- group number 2 (Active Comparator): Group II will will enroll twenty females with PCOS and Psoriasis who will follow low calorie diet and daily metformin for 12 weeks
  Interventions: Behavioral: diet restriction

INTERVENTIONS:
Behavioral: exercise and diet restriction — Group I will enroll twenty females with PCOS and Psoriasis who will apply forty minutes walking on treadmill three times per week for 12 weeks. Also Group I will follow low calorie diet and daily metformin for 12 weeks.
  Arms: group number 1
Behavioral: diet restriction — Group II will will enroll twenty females with PCOS and Psoriasis who will follow low calorie diet and daily metformin for 12 weeks
  Arms: group number 2

SUMMARY:
Women with psoriasis usually develop many complications including polysyctic ovarian syndrome (PCOS). Nowdays, diet restriction combimed with phsyical exercises may improve both problems

DETAILED DESCRIPTION:
Forty Women with psoriasis with PCOS will be enrolled to be catogrized to Group I or group II. Group I will enroll twenty females with PCOS and Psoriasis who will apply forty minutes walking on treadmill three times per week. Also Group I will follow low calorie diet and daily metformin for 12 weeks. Group II will will enroll twenty females with PCOS and Psoriasis who will follow low calorie diet and daily metformin for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* obese (class I) women
* chronic plaque psoriasis
* polyscytic ovarian syndrome

Exclusion Criteria:

* cardiac dysfucntions
* liver diseases
* repsiratory disease
* vascular diseases

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Psoariasis area and severity index | it will be measured after 12 weeks
  is an index used to express the severity of psoriasis. It combines the severity (erythema, induration and desquamation) and percentage of affected area

SECONDARY OUTCOMES:
body mass index | It will be measured after 12 weeks
  it will be assessed after emptying bladder and bowel
waist circumference | It will be measured after 12 weeks
  it will be measured at level of ambilicus
waist hip ratio | It will be measured after 12 weeks
  it will be assessed after dividing waist circumference on hip circumference
testesterone | it will be measured after 12 weeks
  it will be assessed in serum
ratio of luteinizing hormone and follicle-stimulating hormone | It will be measured after 12 weeks
  it is anindicator on function of sex hormones
Dehydroepiandrosterone | It will be measured after 12 weeks
  it will be assessed in plasma
Dermatology life Quality Index | It will be measured after 12 weeks
  it assess impact of skin disease on quality of life
insuiln | It will be measured after 12 weeks
  it will be assessed in plasma
fasting blood glucose | It will be measured after 12 weeks
  it will be assessed in plasma
HOMA-IR | It will be measured after 12 weeks
  Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) is classically considered to be a good insulin resistance (IR) index
triglycerides | It will be measured after 12 weeks
  it will be assessed in plasma
total cholesterol | It will be measured after 12 weeks
  it will be assessed in plasma
high density lipoprotein | It will be measured after 12 weeks
  it will be assessed in plasma
low density lipoprotein | It will be measured after 12 weeks
  it will be assessed in plasma
systolic blood pressure | It will be measured after 12 weeks
  it will be assessed via manual sphygmmanometer
diatolic blood pressure | It will be measured after 12 weeks
  it will be assessed via manual sphygmmanometer

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Giza, Dokki, Egypt